CLINICAL TRIAL: NCT00298662
Title: A Pilot Safety and Tolerability Open-Label Study of Interferon Beta-1b in Combination With Tacrolimus in Patients Suffering From Multiple Sclerosis Who Have Failed Treatment With Approved Disease Modifying Agents
Brief Title: Combination Therapy of Betaseron-Prograf in Multiple Sclerosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Clinique de sclérose en plaques et neuromusculaire de l'Outaouais (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 137-020826
Record Dates: First submitted 2006-03-02; First posted 2006-03-03 (Estimated); Last update posted 2006-03-03 (Estimated); Status verified 2005-09

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Betaseron-Prograf; patients of Multiple Sclerosis; Secondary Progressive type; Relapsing-Remitting type
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1b; Tacrolimus

INTERVENTIONS:
Drug: Interferon beta-1b and Tacrolimus

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of a combination of interferon beta 1-b (Betaseron®) and tacrolimus (Prograf®) in patients suffering from multiple sclerosis (MS) who have failed treatment with currently approved drugs for MS

Prograf is an immunosuppressant that weakens the immune reactions responsible to protect the organism against infections. It is currently available on the market for patients who have received an organ transplant, to prevent rejection. Because of its effect on the immune system, theoretically, Prograf should exert a significant effect in MS. It has been tried in a small number of MS patients at a lower dose than the one used in organ transplant, however the results of the study did not allow to draw definite conclusions on its safety and efficacy in MS.

Betaseron is approved in Canada for the reduction of the frequency of relapses in patients with relapsing-remitting MS and for the slowing of progression and reduction of the frequency of relapses in patients with secondary-progressive MS. The combination of Betaseron and Prograf may result in an additive effect or an increase in the actions of the drugs. However, the combination of the two drugs has never been studied.

The aim of this study is to see how well the combination of Betaseron and Prograf is tolerated by patients with MS. The side effects of the treatment, if any, will be followed. In addition, the efficacy of the combination will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* relapsing-remitting or secondary-progressive multiple sclerosis
* patients who have failed treatment with approved immunomodulator drugs (having experienced same or higher annual relapse rate or having experinced progression on the EDSS scale)
* Expanded Disability Status Scale (EDSS) score less than 7.0

Exclusion Criteria:

* any of the following conditions: diabetes mellitus, uncontrolled hypertension, active infection or viral diseases

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30
Dates: Start 2003-02; Study Completion 2006-09

PRIMARY OUTCOMES:
safety and tolerability
relapse rate
number of T2 godolinium enhencing lesions on MRI
expanded disease severity score (EDSS)
multiple sclerosis functional composite(MSFC)

CONTACTS AND LOCATIONS:
Overall Officials: François Jacques, Principal Investigator — Multiple Sclerosis Clinic - Hull Hospital
Locations (1):
- Clinique de sclérose en plaques et neuromusculaire, Gatineau, Quebec, Canada